CLINICAL TRIAL: NCT05803356
Title: Genetic and Immunologic Characterization of Inborn Errors of Immunity
Brief Title: Genetic and Immunologic Characterization of IEI
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 24/17
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Immunity Disorders; Inborn Errors of Immunity
Keywords: inborn errors of immunity; genotype-phenotype correlation; drugs repositioning; genetics
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inborn Errors of Immunity (IEI) include clinically heterogeneous rare genetic diseases depending on mutations in about 300 different genes. Clinically, this group of diseases is characterized by the presence of infectious, inflammatory, autoimmune, and lymphoproliferative symptoms. Understanding the pathogenesis of these diseases can guide the implementation of targeted therapies and improve prognosis.

In recent years, IEI have been described that do not necessarily present with repeated infectious symptoms but rather with autoimmune, lymphoproliferative, and autoinflammatory manifestations, or with forms of immunodeficiency with a spectrum of susceptibility to one or few infectious agents. In this case, simple laboratory tests are not sufficient to characterize the disease since no particular immunophenotypic changes are evident. To correct classify the patients and to improve knowledge on the pathogenesis of the diseases, complex immunologic-functional studies are required. These studies should be started prior to genetic analysis, with the aim of targeting and narrowing it down. Although the ever-decreasing costs of Next Generation Sequencing (NGS) methods make it convenient to analyse many genes or even the entire exome simultaneously, the analysis of the data resulting from NGS can be complex and provide results of uncertain interpretation. In these cases, immunologic-functional studies can clarify the real causal role of the identified genetic variants.

The identification of genotype-phenotype correlation is crucial to establish new therapeutic targets for diseases orphan of specific etiological treatments. In vitro and in vivo disease models are key tools to test drugs repositioning, as was the case for Lapaquistat in the treatment of periodic fevers caused by de-regulation of the cholesterol metabolic pathway.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected IEI

Exclusion Criteria:

* No consent from the patients' guardians
* Subjects undergoing hematopoietic stem cell transplantation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatrics subjects with suspected Inborn Errors of Immunity
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To identify immunologic-functional characteristics of IEI subjects | Within 30 days of enrollment
  Several test will be carried out on peripheral blood samples (i.e.,evaluation of lymphocyte subpopulations, natural killer cell degranulation assay, intracellular protein expression analysis, interferon signature in real time PCR).
To identify genetic characteristics of IEI subjects | Within 30 days of enrollment
  Using NGS and exome analysis

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Tommasini, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS materno infantile Burlo Garofolo, Trieste, Italy